CLINICAL TRIAL: NCT00683618
Title: A Randomised, Double-blind Trial to Compare the Efficacy of Rosuvastatin 5 and 10 mg to Atorvastatin 10 mg in the Treatment of High Risk Patients With Hypercholesterolemia Followed by an Open Label Treatment Period With Rosuvastatin Up-titrated to the Maximum Dose of 20 mg for Those Patients Who do Not Achieve Goal
Brief Title: Compare the Efficacy of Rosuvastatin to Atorvastatin in High Risk Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D356FC00007
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Hypercholesterolemia
Keywords: HMG-CoA; LDL-C; CHD
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Rosuvastatin 5mg qd
  Interventions: Drug: Rosuvastatin
- 2 (Experimental): Rosuvastatin 10mg qd
  Interventions: Drug: Rosuvastatin
- 3 (Active Comparator): Atorvastatin 10mg qd
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Capsule/Tablet, oral, qd, 6 or 12 weeks
  Other Names: Crestor
  Arms: 1; 2
Drug: Atorvastatin — Capsule/Tablet, 10mg, oral, qd, 6 weeks
  Other Names: Lipitor
  Arms: 3

SUMMARY:
This trial is to compare the efficacy, safety and tolerability of Rosuvastatin with Atorvastatin by assessing the change of LDL-C in patients with hypercholesterolemia and history of coronary heart disease (CHD) or risk equivalent, or a 10 year CHD risk of no less than 10%, following 6-week treatment and a possible 6 week extension treatment.

ELIGIBILITY:
Inclusion Criteria:

* Treated for or diagnosed hypercholesterolemia or have had a high risk with hypercholesterolemia
* LDL-C between 3.36mmol/L and 6.5 mmol/L if not treated with statin or between 2.6mmol/L and 4.14 mmol/L
* Fasting triglyceride less than 4.52mmol/L

Exclusion Criteria:

* History of statin induced myopathy
* Unstable or uncontrolled cardiovascular diseases
* Familial dysbetalipoproteinemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 934 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Eckerd, Study Director — AZ Pharmaceuticals - US; Zhao Shuiping, Principal Investigator — 2nd hospital of Xiangya medical university
Locations (6):
- China (6):
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Shenyang, Liaoning
  - Research Site, Beijing
  - Research Site, Shanghai
  - Research Site, Tianjin

REFERENCES:
- [Derived] Zhao S, Peng D. Efficacy and safety of rosuvastatin versus atorvastatin in high-risk Chinese patients with hypercholesterolemia: a randomized, double-blind, active-controlled study. Curr Med Res Opin. 2018 Feb;34(2):227-235. doi: 10.1080/03007995.2017.1371584. Epub 2017 Sep 18. PMID 28836458

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total 934 patients were enrolled to the study, the study was conducted at 13 investigational sites in China. The first patient was enrolled on 27 May 2008, the last patient was completed on 16 Jul 2009.
Pre-assignment Details: There is a dietary lead in period before randomization. 934 patients started the dietary lead in period. 436 patients completed this period. The baseline measurement is based on the ITT population. Patients included in ITT population in each arm is : Rosuvastatin 5mg 136, Rosuvastatin 10mg 139 and Atorvastatin 10mg 139.
Groups:
- Rosuvastatin 5mg; Rosuvastatin 10mg; Atorvastatin 10mg: Taken orally once daily
Period: Randomised Treatment Period
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Started | 145 | 145 | 146
Completed | 139 | 143 | 140
Not Completed | 6 | 2 | 6
Not completed — Withdrawal by Subject | 4 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 2
Not completed — Reason not provided | 0 | 0 | 2
Period: Extension Treatment Period
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Started | 36 | 23 | 0
Completed | 33 | 23 | 0
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg | Total
Number analyzed (Participants) | 136 | 139 | 139 | 414
Age Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (8.51) | 59.7 (10.57) | 58.4 (9.29) | 59.5 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 85 | 77 | 246
  Male | 52 | 54 | 62 | 168
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 136 | 139 | 139 | 414
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
  Nativ Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
Low density lipoprotein cholesterol (LDL-C level) [Mean (Standard Deviation); unit: mmol/L] | 4.242 (0.6769) | 4.131 (0.6818) | 4.213 (0.6617) | 4.186 (0.6717)
triglyceride (TG) level [Mean (Standard Deviation); unit: mmol/L] | 1.921 (0.7825) | 2.042 (0.9164) | 2.061 (0.8971) | 1.991 (0.8494)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) Concentration After 6 Weeks of Treatment Comparing Rosuvastatin 5mg With Atorvastatin 10mg
Description: Analyzed with analysis of covariance (ANCOVA) model with factors fitted for treatment, centre, risk factor, lipid concentration at baseline, treatment by centre and treatment by risk factor with a two-sided significance level of 0.025 on ITT population.
Time Frame: baseline, 6 weeks
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 5mg | Atorvastatin 10mg
Number analyzed (Participants) | 136 | 139
percent change | -41.70 (2.62) [lower limit 2.62] | -38.67 (2.64) [lower limit 2.64]

2. Primary Outcome: Percentage Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) Concentration After 6 Weeks of Treatment Comparing Rosuvastatin 10mg With Atorvastatin 10mg
Description: Analyzed with analysis of covariance (ANCOVA) model with factors fitted for treatment, centre, risk factor, lipid concentration at baseline, treatment by centre and treatment by risk factor with a significance level of 0.025 on ITT population.
Time Frame: baseline, 6 weeks
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 139 | 139
Percent change | -46.28 (2.62) [lower limit 2.62] | -38.67 (2.64) [lower limit 2.64]

3. Secondary Outcome: Percentage Change From Baseline in High Density Lipoprotein-Cholesterol (HDL-C) at Week 6
Description: Analyzed with analysis of covariance (ANCOVA) model with factors fitted for treatment, centre, risk factor, lipid concentration at baseline, treatment by centre and treatment by risk factor with a significance level of 0.05 on ITT population.
Time Frame: baseline, 6 weeks
Population: Patients who have baseline HDL-C and at least one post baseline HDL-C. Not all patients in ITT meet the conditions since ITT is for all lipid variables instead of individual variable.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 134 | 137 | 135
percent change | 5.63 (2.29) [lower limit 2.29] | 6.82 (2.29) [lower limit 2.29] | 3.64 (2.31) [lower limit 2.31]

4. Secondary Outcome: Percentage Change From Baseline in Total Cholesterol (TC ) at Week 6
Description: as for outcome 3
Time Frame: baseline, 6 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 135 | 139 | 139
percent change | -29.62 (1.92) [lower limit 1.92] | -33.14 (1.91) [lower limit 1.91] | -28.06 (1.93) [lower limit 1.93]

5. Secondary Outcome: Percentage Change From Baseline in Triglycerides (TG) at Week 6
Description: as for outcome 3
Time Frame: baseline, 6 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 135 | 139 | 139
Percent change | -20.09 (4.72) [lower limit 4.72] | -22.05 (4.69) [lower limit 4.69] | -20.67 (4.73) [lower limit 4.73]

6. Secondary Outcome: Percentage Change From Baseline in Non High Density Lipoprotein-Cholesterol (nonHDL-C) at Week 6
Description: as for outcome 3
Time Frame: baseline, 6 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 134 | 137 | 134
percent change | -38.60 (3.57) [lower limit 3.57] | -46.08 (3.57) [lower limit 3.57] | -38.50 (3.60) [lower limit 3.60]

7. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein B (ApoB) at Week 6
Description: as for outcome 3
Time Frame: baseline, 6 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 134 | 139 | 139
percent change | -36.55 (2.40) [lower limit 2.40] | -41.21 (2.40) [lower limit 2.40] | -34.67 (2.41) [lower limit 2.41]

8. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein A-I (ApoA-I) at Week 6
Description: as for outcome 3
Time Frame: baseline, 6 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 134 | 139 | 139
percent change | 3.67 (1.99) [lower limit 1.99] | 4.25 (1.98) [lower limit 1.98] | 1.79 (2.00) [lower limit 2.00]

9. Secondary Outcome: Percentage Change From Baseline in Total Cholesterol/High Density Lipoprotein-Cholesterol (TC/HDL-C) at Week 6
Description: as for outcome 3
Time Frame: baseline, 6 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 134 | 137 | 134
percent change | -32.95 (2.96) [lower limit 2.96] | -38.04 (2.96) [lower limit 2.96] | -31.92 (2.99) [lower limit 2.99]

10. Secondary Outcome: Percentage Change From Baseline in Low Density Lipoprotein Cholesterol/High Density Lipoprotein Cholesterol (LDL-C/HDL-C) at Week 6
Description: as for outcome 3
Time Frame: baseline, 6 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 134 | 137 | 134
percent change | -44.07 (3.17) [lower limit 3.17] | -50.27 (3.16) [lower limit 3.16] | -41.04 (3.19) [lower limit 3.19]

11. Secondary Outcome: Percentage Change From Baseline in Non High Density Lipoprotein Cholesterol/High Density Lipoprotein Cholesterol (nonHDL-C/HDL-C) at Week 6
Description: as for outcome 3
Time Frame: baseline, 6 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 134 | 137 | 134
percent change | -41.79 (11.54) [lower limit 11.54] | -56.63 (11.52) [lower limit 11.52] | -48.33 (11.64) [lower limit 11.64]

12. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein B/Apolipoprotein A I (ApoB/ApoA-I) at Week 6
Description: as for outcome 3
Time Frame: baseline, 6 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 134 | 139 | 139
percent change | -37.62 (3.15) [lower limit 3.15] | -41.87 (3.14) [lower limit 3.14] | -35.15 (3.16) [lower limit 3.16]

13. Secondary Outcome: Percentage of Patients Achieved ATP III Guideline (2001) Low Density Lipoprotein Cholesterol (LDL-C) Goal at Week 6
Description: The percentage of patients achieved LDL-C goal is done in ITT population.
  National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) guideline (2001) LDL-C goal:
  Moderately high risk: 2+ risk factors (10-year risk 10%-20%): LDL-C goal < 3.36mmol/L(130mg/dL), non-HDL-C goal < 4.14mmol/L (160mg/dL) ; High risk: Coronary Heart Disease (CHD) or CHD risk equivalents (10-year risk >20%): LDL-C goal< 2.60mmol/L (100mg/dL), non-HDL-C goal < 3.36mmol/L (130mg/dL)
Time Frame: week 6
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 136 | 139 | 139
percentage of patients | 61.0 | 79.1 | 58.3

14. Secondary Outcome: 6 weeksPercentage of Patients Achieved ATP III Guideline (2001) Non High Density Lipoprotein-Cholesterol (nonHDL-C) Goal at Week 6
Description: The percentage of patients achieved LDL-C goal is done in ITT population.
  National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) guideline (2001) LDL-C goal:
  Moderately high risk: 2+ risk factors (10-year risk 10%-20%): LDL-C goal < 3.36mmol/L(130mg/dL); non-HDL-C goal < 4.14mmol/L (160mg/dL) ; High risk: Coronary Heart Disease (CHD) or CHD risk equivalents (10-year risk >20%): LDL-C goal< 2.60mmol/L (100mg/dL),non-HDL-C goal < 3.36mmol/L (130mg/dL)
Time Frame: week 6
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 136 | 139 | 139
percentage of patients | 66.9 | 78.4 | 60.4

15. Secondary Outcome: Percentage of Patients Achieved National Cholesterol Education Program Adult Treatment Panel (NCEP ATP) III Guideline (2001) Low Density Lipoprotein-Cholesterol (LDL-C) Goal After Titration
Description: as for outcome 13
Time Frame: from week 6 to week 12
Population: Patients did not achieve NCEP ATP III LDL-C goal at the end of 6 weeks randomised treatment period, they entered into extension treatment period upon investigator's discretion.
Measure: Number; unit: percentage of patients
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Number analyzed (Participants) | 34 | 21 | 0
percentage of patients | 41.2 | 47.6 |

ADVERSE EVENTS:
Arm/Group | Rosuvastatin 5mg | Rosuvastatin 10mg | Atorvastatin 10mg
Serious Adverse Events (participants affected / at risk) | 1/145 | 0/145 | 1/146
Other Adverse Events (participants affected / at risk) | 5/145 | 3/145 | 0/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 5mg (N=145) | Rosuvastatin 10mg (N=145) | Atorvastatin 10mg (N=146)
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 5mg (N=145) | Rosuvastatin 10mg (N=145) | Atorvastatin 10mg (N=146)
Alanine Aminotransferase (Investigations) | 2 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 2 | 3 | 0
Myalgia (Renal and urinary disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No